CLINICAL TRIAL: NCT03658811
Title: Evaluation of the Safety and Efficacy of Intense Pulse Light Treatment With Meibomian Gland Expression of Upper Eyelids for Dry Eye Disease
Brief Title: Intense Pulse Light Treatment With Meibomian Gland Expression of the Upper Eyelids in Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toyos Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCLum-001
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2018-12

CONDITIONS: Dry Eye
Keywords: meibomian gland dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Intervention Model Description: Patient were enrolled in the study if they had visible signs of upper lid meibomian gland dysfunction and persistent dry eye symptoms and pain despite treatment with conservative dry eye therapies.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Upper eyelid meibomian gland dysfunction (Experimental): Patients with symptoms of dry eye disease in spite of previous or current use of currently available over the counter or prescription medications for dry eye and evidence of upper eyelid meibomian gland dysfunction and no prior intense pulsed light treatments or meibomian gland expression treatments
  Interventions: Device: intense pulsed light

INTERVENTIONS:
Device: intense pulsed light — Use of 6 mm SapphireCool light guide to treat upper lid margins from tragus to tragus including the nose

SUMMARY:
Upper eyelid treatment has not been used with previously described methods of treatment of dry eye disease using intense pulsed light therapy because the upper lids disease was typically not as advanced as lower lid and because direct treatment of the upper lid was not felt to be necessary as each light pulse extended over the entire periorbita even when concentrated on the lower lid.

DETAILED DESCRIPTION:
Dry eye disease is an under-diagnosed and growing problem. Intense pulsed light has been a proven method of improving the signs and symptoms of meibomian gland dysfunction including lid margin vascularity, meibum viscosity, OSDI mean score and tear break up. This study looks at the safety and effect of treatment of upper lids only to evaluate the safety and efficacy of direct upper lid treatment on the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* subjects older than 18
* cloudy or inspissated meibomian glands in both upper lids
* ocular pain due to dry eye unrelieved by current or prior use of conservative topical dry eye medications including but not limited to over the counter artificial tears, lifitegrast, cyclosporine, or sodium chloride.

Exclusion Criteria:

* Patients with eyelid abnormalities
* intense pulsed light treatment within the past year.
* Patients on oral retinoids,
* patients undergoing intraocular surgery within the past year,
* patients with uncontrolled ocular disease,
* Fitzpatrick skin type V or VI,
* neuro-paralysis in the planned treatment area in the past 6 months,
* pre-cancerous lesions in the planned treatment area.
* New topical eye treatments,
* previous expression of meibomian glands,
* legally blind in one eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Toyos Clinic, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
Excel spreadsheet with data but no identifying characteristics could be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Upper Eyelid Meibomian Gland Dysfunction
Started | 19
Completed | 16
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Upper Eyelid Meibomian Gland Dysfunction
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 64.05 [49 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Non-invasive Tear Break up Time (TBUT)
Description: average of 3 measurements (in seconds) using fluorescein dye and stopwatch to monitor first sign of tear film break up
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Upper Eyelid Meibomian Gland Dysfunction
Number analyzed (Participants) | 19
seconds
  TBUT OD (right eye) | 3.9 [2.6 to 5.3]
  TBUT OS (left eye) | 4.0 [2.6 to 5.4]

2. Secondary Outcome: Measure of Visual Analog Scale Pain Over Last 24 Hours
Description: measure (in millimeters) of pain on scale of minimum of 0 mm(no pain)- maximum of 100mm (maximal pain and worse outcome)
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Upper Eyelid Meibomian Gland Dysfunction
Number analyzed (Participants) | 19
millimeters | 65.42 (0.01)

3. Secondary Outcome: Ocular Discomfort Frequency Assessment on Visual Analog Scale
Description: scale of minimum of 0 mm (no episodes)-maximum of 100 mm (constant painful episodes and worse outcome) frequency of dry eye pain episodes
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Upper Eyelid Meibomian Gland Dysfunction
Number analyzed (Participants) | 19
millimeters | 28.27 (0.01)

4. Secondary Outcome: Measure of Visual Analog Scale Pain
Description: measure of pain since last visit on scale of minimum of 0 mm (no pain)- maximum of 100 mm (maximal pain and worse outcome)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Upper Eyelid Meibomian Gland Dysfunction
Number analyzed (Participants) | 19
millimeters | 26.93 (0.01)

ADVERSE EVENTS:
Time Frame: Adverse events were noted during patients enrollment in the study, at minimum 8 weeks and at most 16 weeks.
Arm/Group | Upper Eyelid Meibomian Gland Dysfunction
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 13/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Upper Eyelid Meibomian Gland Dysfunction (N=19)
Mild Stinging (Eye disorders) | 5 (5) — Mild stinging from the light therapy on the upper eyelid
Moderate discomfort (Eye disorders) | 13 (13) — Mild discomfort during digital Expression of upper eyelid

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT03658811/Prot_SAP_000.pdf